CLINICAL TRIAL: NCT05066789
Title: Comparison of Polymer-Free Cobalt-Chromium Thin Drug-Coated Stents With Biodegradable Polymer Ultrathin Sirolimus-Eluting Stents and Prasugrel Monotherapy With Conventional 12-Month Dual Antiplatelet Therapy
Brief Title: CHoice of Optimal Anti-Thrombotic Strategy in Patients Undergoing Implantation of Coronary Drug-Eluting Stents 4
Acronym: SMART-CHOICE4
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Ending early registration due to low registration status and lack of research
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joo-Yong Hahn, Professor, Samsung Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CHOICE-4
Record Dates: First submitted 2021-09-15; First posted 2021-10-04 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; Acute coronary syndrome; Antiplatelet Therapy; Drug eluting stent
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: multi-center, open label, two-by-two factorial, randomized, noninferiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Biodegradable Polymer DES (Active Comparator): Patients will be randomized to either the polymer-free drug-coated stent (DCS) group or the biodegradable polymer drug-eluting (DES) group with 1:1 ratio.
  This group will use Orsiro Mission stent during the index procedure.
  Interventions: Device: Type of stent
- 12-month DAPT (Active Comparator): Patients will be randomized to either the prasugrel monotherapy group or the 12-month dual antiplatelet therapy (DAPT) group with 1:1 ratio unless patients have additional exclusion criteria for antiplatelet study.
  This group will receive 12-month DAPT of aspirin (100mg once daily) plus prasugrel (10mg once daily).
  Interventions: Drug: Duration of DAPT
- Polymer-free DCS (Experimental): Patients will be randomized to either the polymer-free drug-coated stent (DCS) group or the biodegradable polymer drug-eluting (DES) group with 1:1 ratio.
  This group will use BioFreedom Ultra stent during the index procedure.
  Interventions: Device: Type of stent
- Prasugrel monotherapy (Experimental): Patients will be randomized to either the prasugrel monotherapy group or the 12-month dual antiplatelet therapy (DAPT) group with 1:1 ratio unless patients have additional exclusion criteria for antiplatelet study.
  This group will receive aspirin (100mg once daily) plus prasugrel (10mg once daily) for 1 month and thereafter prasugrel (10mg once daily) alone.
  Interventions: Drug: Duration of DAPT

INTERVENTIONS:
Device: Type of stent — 1:1 randomization to biodegradable polymer DES (Orsiro Mission) and polymer-free DCS (Biofreedom)
  Arms: Biodegradable Polymer DES; Polymer-free DCS
Drug: Duration of DAPT — 1:1 randomization to 1-month DAPT thereafter prasugrel monotherapy and 12-month DAPT (aspirin + prasugrel)
  Arms: 12-month DAPT; Prasugrel monotherapy

SUMMARY:
This study is multi-center, open label, two-by-two factorial, randomized, noninferiority trial to compare the efficacy and safety of polymer-free cobalt-chromium thin drug-coated stents (BioFreedom Ultra) with biodegradable polymer ultrathin sirolimus-eluting stents (Orsiro Mission) and prasugrel monotherapy after 1-month dual antiplatelet therapy (DAPT) of aspirin plus prasugrel with 12-month DAPT of aspirin plus prasugrel in patients with acute coronary syndrome undergoing percutaneous coronary intervention.

DETAILED DESCRIPTION:
Polymer is the key component of drug-eluting stents (DES) for facilitation of drug loading and control of drug release. However, durable polymer of the 1st generation DES has been considered to induce inflammation and to be associated with fatal complications such as very late stent thrombosis. To overcome this shortcoming, biodegradable polymer has been applied to the DES system. In several head-to-head comparison, ultrathin strut biodegradable polymer sirolimus-eluting Orsiro stent demonstrated comparable or superior outcomes compared with durable polymer everolimus-eluting stents. As a result, Orsiro stent is considered one of the standard contemporary DESs.

On the other hand, polymer-free drug-coated stents (DCS) have been developed as an alternative to durable and biodegradable polymer DES. The biolimus A9-coated BioFreedom stent is the representative polymer-free drug-coated stent and was superior to a bare-metal stent in patients treated with 1-month dual antiplatelet therapy (DAPT). However, it failed to show noninferiority for major adverse cardiovascular events at 12 months when compared with the ultrathin strut biodegradable polymer sirolimus-eluting Orsiro stent in an all-comers population, mainly due to increased target lesion revascularization (TLR). On top of possible insufficient or uncontrolled drug delivery at stented site due to absence of a drug carrier, thick strut (112 µm) and stainless steel alloy may explain a higher rate of TLR in the BioFreedom stent group compared with the Orsiro stent group. The BioFreedom Ultra stent is a novel cobalt-chromium thin stent (84 µm) with biolimus A9-coating. With advancement in stent alloy and strut thickness, treatment efficacy and safety of the BioFreedom Ultra stent would be comparable to the new version of Orsiro stent (Orsiro Mission) among patients with acute coronary syndrome (ACS).

Patients with ACS undergoing percutaneous coronary intervention (PCI) with DES are currently recommended to use 12 months of DAPT, consisting of aspirin and P2Y12 inhibitor. Although use of DAPT reduces ischemic events, including stent thrombosis, bleeding events increase in return. Hence, considering the aforementioned advancement of stent devices, shorter duration of DAPT and switching to a potent P2Y12 inhibitor monotherapy would be possible. This has been demonstrated in several recent studies. However, although prasugrel was superior to ticagrelor in lowering ischemic events, these studies mainly used ticagrelor as a solely used antiplatelet agent, and studies verifying the effect of prasugrel monotherapy after short duration of DAPT are limited to date. In addition, in these studies, DAPT was maintained for mostly at least 3 months in the ACS situation. With advancement of devices, duration of DAPT may be further reduced. In other words, prasugrel monotherapy after 1 month of DAPT of aspirin plus prasugrel would be comparable to 12-month DAPT of aspirin plus prasugrel.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 19 years of age
2. Subject who is able to understand risks, benefits and treatment alternatives and sign informed consent voluntarily.
3. Patients presenting with ACS (ST-elevation myocardial infarction [STEMI], non-ST-elevation myocardial infarction [NSTEMI], or unstable angina)
4. Patients with at least one lesion with equal or greater than 50% diameter stenosis requiring treatment with drug-eluting stents (DES) in native coronary artery or graft

Exclusion Criteria:

1. Patients unable to provide consent
2. Patients with known intolerance to aspirin, clopidogrel, prasugrel, or major components of drug-eluting stents
3. Patients who have non-cardiac co-morbid conditions with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment)
4. Patients who need chronic anti-coagulation therapy
5. Patients with active pathological bleeding
6. Pregnant or lactating women

Additional Exclusion Criteria for Antiplatelet Comparison Study:

1. Patients with history of stroke or transient ischemic attack
2. Patients 75 years of age or older
3. Patients weighing less than 60 kg

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Stent Comparison Study: target-lesion failure (TLF) | 1 year
  a composite of cardiac death, target vessel-myocardial infarction, or clinically indicated target-lesion revascularization by percutaneous or surgical methods
Antiplatelet Comparison Study: net adverse clinical events (NACE) | 1 year
  a composite of major adverse cardiac and cerebrovascular events (MACCE) and clinically relevant bleeding

SECONDARY OUTCOMES:
Stent Comparison Study: TLF | 3 years
  a composite of cardiac death, target vessel-myocardial infarction, or clinically indicated target-lesion revascularization by percutaneous or surgical methods
Stent Comparison Study: target-vessel failure | 1 and 3 years
  a composite of cardiac death, target vessel-MI, or clinically indicated target-vessel revascularization by percutaneous or surgical methods
Stent Comparison Study: cardiac death | 1 and 3 years
  cardiac death
Stent Comparison Study: target-vessel myocardial infarction (MI) | 1 and 3 years
  target-vessel MI
Stent Comparison Study: clinically indicated TLR | 1 and 3 years
  clinically indicated TLR
Stent Comparison Study: stent thrombosis | 1 and 3 years
  definite or probable by Academic Research Consortium [ARC] definition
Stent Comparison Study: clinically indicated target-vessel revascularization (TVR) | 1 and 3 years
  clinically indicated target-vessel revascularization (TVR)
Stent Comparison Study: cardiac death or MI | 1 and 3 years
  cardiac death or MI
Stent Comparison Study: cardiac death, MI, or stent thrombosis | 1 and 3 years
  cardiac death, MI, or stent thrombosis
Stent Comparison Study: all-cause death | 1 and 3 years
  all-cause death
Stent Comparison Study: MI | 1 and 3 years
  MI
Stent Comparison Study: all-cause death or MI | 1 and 3 years
  all-cause death or MI
Stent Comparison Study: any revascularization | 1 and 3 years
  any revascularization
Stent Comparison Study: restricted mean survival time for the TLF | 1 and 3 years
  restricted mean survival time for the TLF
Antiplatelet Comparison Study: MACCE | 1 year
  a composite of all-cause death, MI, and stroke
Antiplatelet Comparison Study: clinically relevant bleeding | 1 year
  bleeding Academic Research Consortium (BARC) type 2, 3 or 5 bleeding
Antiplatelet Comparison Study: all-cause death | 1 year
  all-cause death
Antiplatelet Comparison Study: MI | 1 year
  MI
Antiplatelet Comparison Study: stroke | 1 year
  stroke
Antiplatelet Comparison Study: cardiac death | 1 year
  cardiac death
Antiplatelet Comparison Study: stent thrombosis | 1 year
  definite or probable by ARC definition
Antiplatelet Comparison Study: all-cause death or MI | 1 year
  all-cause death or MI
Antiplatelet Comparison Study: cardiac death or MI | 1 year
  cardiac death or MI
Antiplatelet Comparison Study: cardiac death, MI, or stent thrombosis | 1 year
  cardiac death, MI, or stent thrombosis
Antiplatelet Comparison Study: BARC type 3 or 5 bleeding | 1 year
  BARC type 3 or 5 bleeding
Antiplatelet Comparison Study: restricted mean survival time for the NACE | 1 year
  restricted mean survival time for the NACE

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Yong Hahn, MD, PhD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No